CLINICAL TRIAL: NCT02547753
Title: Clinical Outcome of Dental Extractions Among Renal Transplant Recipients
Brief Title: Dental Extractions Among Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other); Hospital do Rim e Hipertensão (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marina Helena Cury Gallottini, Full Prof Oral Pathology, University of Sao Paulo
Other Study IDs: CAAE: 45413015.0.0000.0075
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Immunosuppression
Keywords: Tooth extraction; Antibiotic prophylaxis; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and saliva - laboratorial tests
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Transplanted group: patients who are kidney receptors for at least 6 months and need tooth extraction
- Control group: healthy patients who need tooth extraction

SUMMARY:
The literature is rich in studies that explore the type and frequency of oral abnormalities in transplanted recipients, but it is scarce in studies that provide scientific evidence on the risk of complications after invasive interventions on those patients. Within this context, the aim of our study is to evaluate the post-exodontic socket healing in renal transplant recipients compared to a control group and see if some indicators in the population of transplanted people, such complete blood count, serum concentration of immunosuppressive drugs, can help to provide for the host response face a invasive procedures. Therefore, 45 kidney transplant recipients over six months and at least 45 healthy non immunosuppressed adults will be submitted to a maximum of 4 simple dental extractions, always by the same surgeon. Laboratory tests will be performed preoperatively and include: blood count and coagulation - for both groups - and urea, creatinine and serum levels of immunosuppressive drug - only for the study group. Researchers will evaluate the patient in the postoperative 3, 7, 21, and 60 days. The presence, or absence, of post-operative complication and delayed, or not, socket healing will be the results of interest in this study and will be compared between the groups. The data will be evaluated by Pearson's chi-square, Fisher's exact test, Mann-Whitney test, student's T-test and binomial test.

DETAILED DESCRIPTION:
Investigators did not found scientific evidences neither evidence-based research, which support the idea that stable kidney recipients have increased risk for delayed socket repair and wound healing after exodontia or that infections resulted by oral surgery are more common in these patients, despite the drug-induced immunosuppression which they use.

Since there is no scientific evidence about the increased risk of post-exodontic infection, not even about a disorder on the alveolar repair chronology, after exodontia performed in kidney recipients, the aim of our study will be prospectively observe kidney recipients who are undergoing dental extractions.

This prospective cohort study will involve 45 adult kidney recipients for at least 6 months, and 61 non-transplanted and healthy control adults, who need simple extraction of an erupted tooth.

All the patients must be evaluated in the preoperative phase through anamnesis (e.g. collecting data concerning on base diseases, personal history, presence of drug allergy, medications in use, habits and addictions), extra-oral and intra-oral physical examinations and laboratory tests.

Participants must sign the Inform and Clarified Consent Term to participate. Will be disqualified participants that: used antibiotics in the month preceding the extraction, made bisphosphonate therapy, user of illicit drugs, chronic alcoholics, who present with dental emergencies, acute dental or periodontal infections, and patients with cognitive impairment.

One week before the dental extraction will be collected 15ml of blood from participants of both group to perform complete blood count, coagulation tests, urea and creatinine measurements. The serum measurement of the immunosuppressed drug will be performed only in the individuals of study group.

Dental extractions, from one to three erupted teeth, will be performed by the same dentist, specialist in Oral and Maxillofacial Surgery, enabled by the Federal Council of Dentistry, on the ambulatory of CAPE (special care center) , under local anesthesia following the standards described by Peterson et al (2003). The local anesthetic used in all individuals will be prilocaine with epinephrine as vasoconstrictor. After the anesthetic blockade, incision and mucosal detachment, luxation with elevators and tooth removal with forceps will be performed. The surgical technique will be modified according the condition of the tooth on the socket; when necessary tooth sectioning and/or ostectomy will be performed. By the end, curettage of the socket, post-extraction alveolar compression to reduce the width of the same and simple suture with 4.0 silk thread will be carried out.

Each tooth characteristics and each surgery data will be recorded and will include: surgical duration (from the anesthesia to the suture), surgical technique variations, such the use of elevators, forceps, mucoperiosteal flaps, tooth sectioning and/or ostectomy and intraligamentary anesthesia, and number of anesthetics cartridges used.

After the surgery, the patient will press a gauze for 30 minutes in the extraction's region in order to control bleeding. It will be prescribed 750 mg of Acetominophen, up to 3 times a day, for 24 hours. In case of necessity of change in the postoperative therapeutic due to surgical technique variations, data will be recorded and included.

Clinical assessment of healing will be performed by a blinded examiner on 3, 7, 21 and 60 days after surgery. In these periods, the region will always be examined by the same examiner.

Radiographic evaluation will be done with standardized periapical radiographs, with individualized positioners, made in the immediately and 60 days postoperative, which bone density and alveolar crest remodeling will be evaluated by a blinded examiner.

With 21 days postoperative, the socket will be classified as: 1) without complication; or 2) with complications. According to Cheung et al (2001), the following situations will be considered as post-exodontics complications:

Acute alveolar infection (dry socket, fibrinolytic osteitis, alveolar osteitis) or surrounding tissue infection Acute alveolar inflammation.

In case of postoperatively infection, copious irrigation with sodium chloride solution (NaCl 0,9%) will be performed and will be prescribed amoxicilline 500 mg every 8 hours for 7 days and anti-inflammatory nimesulide 100 mg every 12 hours for 5 days. In case of allergy to penicillin, clindamycin will be prescribed at a dose of 300 mg every 8 hours for 7 days.

The second outcome of interest in this study will be observe the total alveolar epithelialization. According to the literature, at 3 days postoperative, the socket is filled with blood clot and fibrin; at 7 days, the socket is filled with granulation tissue; and from 21 days the surgical wound is fully epithelialized. Delayed epithelialization will be considered in case at on the day 21, the socket would not yet fully covered by epithelialized mucosa.

Finally, the third point will be the bone deposition in the socket, at 60 days postoperative.

All data will be transferred to an Excel spreadsheet and analyzed descriptively and associated with each other. Complications will be compared between the two groups. In addition, in the study group, researchers will investigate the occurrence of complications associated with transplantation time, immunosuppressive dose, and presence of comorbidity, such as diabetes.

Exact Fisher's test or Fisher's exact test will be applied, Mann-Whitney's test or Student's T-test and binomial test using the R software, version 2.15.3 (R Development Core Team, 2012). The significance level will be set at 5%. Adjustments to modifying factors such as smoking and presence of diabetes will be analyzed by logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* renal transplantation for more than 6 months

Exclusion Criteria:

* use of antibiotic in the previous month, use of bisphosphonate therapy, use of illicit drugs, chronic use of alcohol, having a dental emergency,having acute dental or periodontal infections, having a cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: kidney transplanted individuals requiring extraction of erupetd teeth
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-10; Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Complication | 21 days
  alveolar healing will be classified in complicated or non-complicated, based on the conditions and symptoms of soft tissue healing

SECONDARY OUTCOMES:
Delayed alveolar healing | 60 days
  alveolar healing will be classified in normal or delayed healing based on the chronology of alveolar and soft tissue healing

CONTACTS AND LOCATIONS:
Overall Officials: Marina Gallottini, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Rubens Caliento, São Paulo, São Paulo
  - University of São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All the data will be available after the end of study
Supporting Information: Study Protocol
Time Frame: Immediately after the end of the study
Access Criteria: General public
URL: https://www.teses.usp.br

REFERENCES:
- [Background] Guggenheimer J, Eghtesad B, Stock DJ. Dental management of the (solid) organ transplant patient. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Apr;95(4):383-9. doi: 10.1067/moe.2003.150. PMID 12686921
- [Background] Brown RS, McIntosh CL, Cotca CC, Glascoe AL. Dental management of a kidney transplant patient. Dent Today. 2012 Jul;31(7):74-6; quiz 78-9. No abstract available. PMID 22891597
- [Background] Byron RJ Jr, Osborne PD. Dental management of liver transplant patients. Gen Dent. 2005 Jan-Feb;53(1):66-9; quiz 70-2. PMID 15779227
- [Background] Cheung LK, Chow LK, Tsang MH, Tung LK. An evaluation of complications following dental extractions using either sterile or clean gloves. Int J Oral Maxillofac Surg. 2001 Dec;30(6):550-4. doi: 10.1054/ijom.2000.0128. PMID 11829239
- [Background] Cohen D, Galbraith C. General health management and long-term care of the renal transplant recipient. Am J Kidney Dis. 2001 Dec;38(6 Suppl 6):S10-24. doi: 10.1053/ajkd.2001.28922. PMID 11729002
- [Background] Georgakopoulou EA, Achtari MD, Afentoulide N. Dental management of patients before and after renal transplantation. Stomatologija. 2011;13(4):107-12. PMID 22362336
- [Background] Guggenheimer J, Mayher D, Eghtesad B. A survey of dental care protocols among US organ transplant centers. Clin Transplant. 2005 Feb;19(1):15-8. doi: 10.1111/j.1399-0012.2005.00251.x. PMID 15659128
- [Background] Hariharan S, Johnson CP, Bresnahan BA, Taranto SE, McIntosh MJ, Stablein D. Improved graft survival after renal transplantation in the United States, 1988 to 1996. N Engl J Med. 2000 Mar 2;342(9):605-12. doi: 10.1056/NEJM200003023420901. PMID 10699159
- [Background] Lockhart PB, Brennan MT, Fox PC, Norton HJ, Jernigan DB, Strausbaugh LJ. Decision-making on the use of antimicrobial prophylaxis for dental procedures: a survey of infectious disease consultants and review. Clin Infect Dis. 2002 Jun 15;34(12):1621-6. doi: 10.1086/340619. Epub 2002 May 23. PMID 12032898
- [Background] Lockhart PB, Loven B, Brennan MT, Fox PC. The evidence base for the efficacy of antibiotic prophylaxis in dental practice. J Am Dent Assoc. 2007 Apr;138(4):458-74; quiz 534-5, 437. doi: 10.14219/jada.archive.2007.0198. PMID 17403736
- [Background] Weinberg MA, Segelnick SL, Kay LB, Nair V. Medical and dental standardization for solid organ transplant recipients. N Y State Dent J. 2013 Nov;79(6):35-40. PMID 24600763
- [Background] Ziebolz D, Hrasky V, Goralczyk A, Hornecker E, Obed A, Mausberg RF. Dental care and oral health in solid organ transplant recipients: a single center cross-sectional study and survey of German transplant centers. Transpl Int. 2011 Dec;24(12):1179-88. doi: 10.1111/j.1432-2277.2011.01325.x. Epub 2011 Sep 8. PMID 21902726
- [Background] Spolidorio LC, Spolidorio DM, Massucato EM, Neppelenbroek KH, Campanha NH, Sanches MH. Oral health in renal transplant recipients administered cyclosporin A or tacrolimus. Oral Dis. 2006 May;12(3):309-14. doi: 10.1111/j.1601-0825.2005.01200.x. PMID 16700742
- [Derived] Caliento R, Sa Fernandes K, Andrade NS, de Santana Sarmento DJ, Pontello Cristelli M, L Ortega K, Gallottini M. Extractions in kidney transplant recipients: A prospective observational pilot study. J Am Dent Assoc. 2022 Mar;153(3):233-240. doi: 10.1016/j.adaj.2021.08.004. Epub 2021 Nov 20. PMID 34794682